CLINICAL TRIAL: NCT04034641
Title: Clinical Study on Bifidobacterium Quadruple Live Bacteria Tablets (Si Lian Kang) Reducing the Incidence Rate of Adverse Reactions in Helicobacter Pylori Quadruple Eradication Therapy and on the Effects of Gastrointestinal Flora
Brief Title: Effect of Probiotics on Helicobacter Pylori Eradication
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Grand Biologic Pharmaceutical, Inc. (Industry)
Collaborators: The First Affiliated Hospital of Nanchang University (Other); The First People's Hospital of Yunnan (Other); Zhejiang Provincial Hospital of TCM (Other); Fifth Affiliated Hospital of Zhengzhou University (Unknown); Nanjing First Hospital, Nanjing Medical University (Other); Xi'an Central Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HangzhouGrand
Record Dates: First submitted 2019-07-22; First posted 2019-07-26 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-07

CONDITIONS: Helicobacter Pylori Eradication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotics plus standard therapy (Experimental)
  Interventions: Drug: Bifidobacterium tetrad live bacteria tablet plus Helicobacter pylori quadruple eradication therapy
- placebo plus standard therapy (Placebo Comparator)
  Interventions: Drug: Bifidobacterium tetrad live bacteria tablet placebo plus Helicobacter pylori quadruple eradication therapy

INTERVENTIONS:
Drug: Bifidobacterium tetrad live bacteria tablet plus Helicobacter pylori quadruple eradication therapy — On day 1-14: Standard therapy: esomeprazole magnesium enteric-coated tablets, amoxicillin granules (A Mo Xian), furazolidone tablets, bismuth potassium citrate granules (Li Zhu De Le) are taken twice a day, once in the morning and once in the evening. Esomeprazole magnesium enteric-coated tablets and bismuth potassium citrate granules (Li Zhu De Le) should be taken 30min before meal; amoxicillin granules (A Mo Xian) and furazolidone tablets should be taken 30min after meal. Probiotic: Bifidobacterium tetrad live bacteria tablets should be taken at noon once a day (30 min after meal ), 9 tablets per time. On day 15-28: Probiotic: Bifidobacterium tetrad live bacteria tablets, taken at noon once a day (30min after meal), 9 tablets per time.
  Arms: probiotics plus standard therapy
Drug: Bifidobacterium tetrad live bacteria tablet placebo plus Helicobacter pylori quadruple eradication therapy — On day 1-14: Standard therapy: esomeprazole magnesium enteric-coated tablets, amoxicillin granules (A Mo Xian), furazolidone tablets, bismuth potassium citrate granules (Li Zhu De Le) are taken twice a day, once in the morning and once in the evening. Esomeprazole magnesium enteric-coated tablets and bismuth potassium citrate granules (Li Zhu De Le) should be taken 30min before meal; amoxicillin granules (A Mo Xian) and furazolidone tablets should be taken 30min after meal. Placebo: Bifidobacterium tetrad live bacteria tablet placebos should be taken at noon once a day ( 30 min after meal ), 9 tablets per time. On day 15-28: Placebo: Bifidobacterium tetrad live bacteria tablet placebos, taken at noon once a day (30min after meal), 9 tablets per time.
  Arms: placebo plus standard therapy

SUMMARY:
The purpose of this clinical trial is to evaluate the clinical efficacy of Bifidobacterium quadruple live bacteria tablets (Si Lian Kang) on reducing the incidence rate of adverse reactions of Helicobacter pylori quadruple eradication therapy and its influence on gastrointestinal flora.

DETAILED DESCRIPTION:
Bismuth agent quadruple therapy (including bismuth agent and proton pump inhibitor combined with two antibiotics) is the first-line strategy to eradicate Helicobacter pylori in China. However, it may cause a series of adverse reactions, such as nausea, diarrhea, abdominal pain, constipation, and abnormal taste, etc., which leads to a decrease in patient compliance, thereby affecting the treatment effect. Many studies have found that adding probiotics to traditional Helicobacter pylori eradication therapies increase eradication rates and reduce the side effects of the treatment. Bifidobacterium tetrad live bacteria tablet is a compound microecological preparation composed of bifidobacterium infantis, lactobacillus acidophilus, enterococcus faecalis and bacillus cereus. This study aims to observe the clinical efficacy of Bifidobacterium quadruple live bacteria tablets (Si Lian Kang) on reducing the incidence rate of adverse reactions in Helicobacter pylori quadruple eradication therapy and on the effects of gastrointestinal flora.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signing the informed consent form;
2. Aged 18-65 years old(including 65), male or female;
3. Patients aged 35-65 years old(including 35) with positive Helicobacter pylori should undergo gastroscopy, and the gastroscopy report shows normal or chronic gastritis;
4. Patients aged 18-35 years (including 18) with positive Helicobacter pylori are not required to perform gastroscopy examination if there is no obvious clinical symptoms, or applying report of gastroscopy within 6 months showing normal or chronic gastritis.

Exclusion Criteria:

1. Gastroscopy report or previous medical history showed significant esophagus-gastric diseases, including gastric cancer, peptic ulcer, oesophagitis and esophageal erosion;
2. Patients with chronic diarrhea and chronic functional constipation;
3. Other systemic diseases, including cardiovascular diseases, lung diseases, liver diseases (transaminase index is more than 2 times higher than the normal value), kidney diseases (creatinine index is higher than the normal value) and other important organs with severe lesions, severe metabolic diseases (diabetes, thyroid diseases), malignant tumors, and severe immune system diseases;
4. Abnormal stool routine results: fecal occult blood (+) or white blood cells (+);
5. Patients with severe psychological or mental diseases;
6. Those with a history of drug abuse or alcohol abuse;
7. Those who are allergic to the drugs in this study;
8. Those who have received Helicobacter pylori eradication therapy;
9. Drugs which affect the intestinal flora(including antibacterial drugs, microecological preparations, intestinal mucosal protectors, Chinese patent medicines, etc.) have been used in the past 1 month or need to be used continuously for more than 1 week in the experiment.
10. Pregnant or lactating women;
11. Participating or after completing other clinical trials Less than 3 months;
12. Others who researchers consider unsuitable for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
the total incidence rate of digestive tract related adverse reactions | baseline, 28 days, 182days
  The patient diary cards (including Bristol stool classification, diarrhea, constipation, abdominal pain, abdominal distension, belching, nausea, vomiting, loss of appetite and changes in taste) are filled in daily from the -14th day to 28th day. The above contents are recorded weekly from the 29th to182th day. to calculate the total incidence rate of digestive tract related adverse reactions mentioned above

SECONDARY OUTCOMES:
the incidence rate of various digestive tract related symptoms | baseline, 28 days, 182days
  to calculate incidence rate of various digestive tract related symptoms including diarrhea, constipation, and other symptoms mentioned above
duration of various digestive tract related symptoms | baseline, 28 days, 182days
  to calculate duration of various digestive tract related symptoms including diarrhea, constipation, and other symptoms mentioned above
stool frequency | baseline, 28 days, 182days
  to evaluate the defecation frequency of diarrhea and constipation
changes in intestinal flora | baseline, 14 days, 28 days, 70 days, 182days
  to evaluate the changes of intestinal flora during the clinical study period
changes in gastric flora | baseline, 70 days
  20 patients are enrolled in the experiment group and control group respectively. Mucosal samples (one gastric antrum and one gastric body) are taken by gastroscopy before treatment. Gastroscope was reexamined 6 weeks after probiotics or placebo withdrawal (the 70th day), and mucosal samples (one gastric antrum and one gastric body) are taken.
Helicobacter pylori eradication rate | 70 days
  to evaluate the results of 13C-urea breath test
adverse events | 28 days,182 days
  Adverse events are assessed during the clinical study period.

CONTACTS AND LOCATIONS:
Overall Officials: Nonghua Lv, master, Principal Investigator — The First Affiliated Hospital of Nanchang University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Xi'an Central Hospital, Xi’an, Shanxi